CLINICAL TRIAL: NCT04509921
Title: Adjustment of Asthma Treatment in Children Based on an Indirect Hyperresponsiveness Test - a Randomized Trial
Brief Title: Adjustment of Asthma Treatment in Children Based on an Indirect Hyperresponsiveness Test
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute for Tuberculosis and Lung Diseases, Poland (Other)
Collaborators: The Regional Public Hospital in Lesko, Poland (Other); University of Rzeszow (Other)
Responsible Party: Principal Investigator, Henryk Mazurek, Clinical Professor; MD, PhD, National Institute for Tuberculosis and Lung Diseases, Poland
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Basic Science
Other Study IDs: BA_BHR
Record Dates: First submitted 2020-08-07; First posted 2020-08-12 (Actual); Last update posted 2020-08-12 (Actual); Status verified 2020-08

CONDITIONS: Asthma in Children
Keywords: asthma; bronchoprovocation; inhaled corticosteroids
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- symptoms group (No Intervention): The asthma treatment adjustments guided by GINA guidelines
- BHR group (Experimental): The asthma treatment adjustments additionally taking account to the results of the bronchial hyperresponsiveness test
  Interventions: Other: asthma treatment adjustment taking account on degree of bronchial hyperresponsiveness

INTERVENTIONS:
Other: asthma treatment adjustment taking account on degree of bronchial hyperresponsiveness — Modification of inhaled corticosteroid dose based on the symptoms and the result of bronchial provocation (BHR group)
  Arms: BHR group

SUMMARY:
The aim of the study is to assess the usefulness of the indirect bronchial hyperresponsiveness test (with hypertonic NaCl) in determining the optimal dose of inhaled steroids to maintain asthma control.

The study was designed as a prospective, real-life, randomized, interventional study. This single-site study is performed at the Allergology Clinic in Lesko.

The study included participants aged 7-15 years who met the eligibility criteria. Eligible participants were selected from a pool of 231 patients with mild asthma, under the care of the Allergology Clinic of the Regional Public Hospital in Lesko (Poland). All participants were diagnosed with chronic mild asthma for at least two years.

Subjects initially enrolled in the study had good asthma control maintained for at least 3 months on low / medium-dose ICS monotherapy, with no exacerbations requiring systemic corticosteroids in the previous 3 months, no respiratory tract infection in last month, and an FEV1 above 80% expected.

Finally, 108 children were enrolled in the study. They were aged 7-15 years, with active mild asthma, confirmed by the presence of bronchial hyperreactivity and symptoms of asthma, emerging after discontinuation of anti-inflammatory treatment.

Participation in the study lasted one year.

The study includes:

4-week run-in period (withdrawal phase) after discontinuation of anti-inflammatory treatment (ICS) with clinical symptoms and medication use recording, completed by the patient and parents.

At the end of this period, spirometry was performed, bronchial hyperreactivity was assessed with the hyperosmolar salt provocation, and the parameters of inflammation were measured: orally exhaled nitric oxide concentration (NO) and peripheral blood eosinophilia. The anti-inflammatory treatment was then resumed (with ICS in the previous doses).

Only patients with active asthma and increased bronchial responsiveness (DRS>0.55) were qualified for the main study. Stratified randomization was performed for age, clinical symptoms, and the degree of bronchial hyperresponsiveness. On this basis, the division into 2 research groups was made:

* a symptom-only monitored treatment group
* a group in which therapy changes were based on the symptoms and degree of bronchial hyperresponsiveness (BHR group).

Patients/parents were provided by an established algorithm for managing asthma symptoms/exacerbations. In the case of loss of asthma control, a beta-agonist was administered (temporarily) and the dose of ICS quadrupled. Patients had the possibility of additional visits - if necessary. Especially, severe exacerbations were verified by the attending physician, and on this basis, oral steroids would be considered.

Throughout the study, the participants kept daily observation charts (clinical symptoms and drug use) and peak expiratory flow rate (PEFR) measurements.

The telephone report was made monthly with the number of days with asthma symptoms and medications used, and this was recorded in the documentation of the study.

The clinical evaluation was performed every 3 months with symptom evaluation, spirometry, exhaled NO, peripheral blood eosinophilia, and BHR measurements (half of the patients).

The treatment adjustments were guided by the patient's and parent's reporting of symptoms, and additionally by the results of periodic clinical assessment (including the assessment of bronchial hyperresponsiveness in the BHR group). This means that the level of treatment intensity (ICS dose) was based on symptom monitoring only in the observation group, and additionally took into account the level of bronchial responsiveness in the BHR monitoring group.

The study was completed after one year of follow-up (4 visits every 3 months). The primary endpoint of the study: the number of asthma exacerbations in both study arms.

Secondary endpoints:

* days with symptoms
* asthma medication days
* final dose of ICS
* spirometry (FEV1, MMEF)
* bronchial hyperreactivity (BHR group only)
* nitric oxide in the exhaled air
* peripheral blood eosinophilia.

ELIGIBILITY:
Inclusion Criteria:

* mild asthma with a stable course of at least 3 months
* good adherence to treatment with low dose ICS

Exclusion Criteria:

* infection or exacerbation of asthma requiring the use of systemic steroids (or changes in the dose of inhaled steroids) in the last 3 months before the study
* other chronic lung diseases or general diseases affecting the respiratory system
* tobacco smoking
* FEV1 below 80% of the predicted value

Ages: 7 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 108 (Actual)
Dates: Start 2018-07-02 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2019-08-30 (Actual)

PRIMARY OUTCOMES:
asthma exacerbations | 12 months
  number of asthma exacerbations

SECONDARY OUTCOMES:
the percentage of participants with asthma exacerbations | 12 months
  the number of patients with at least 1 exacerbation divided by the number of patients in each group
time to the first asthma exacerbation | 12 months
  the median time to the first asthma exacerbation in each group
ICS dose | 12 months
  the final dose of ICS
days with symptoms | 12 months
  total number of days with asthma symptoms
days with asthma medication | 12 months
  total number of days with bronchodilator use
blood eosinophilia | 12 months
  number of blood eosinophils
exhaled nitric oxide | 12 months
  orally exhaled nitric oxide concentration
spirometry | 12 months
  FEV1, forced vital capacity (FVC) and FEF (MMEF) values

CONTACTS AND LOCATIONS:
Locations (1):
- The Regional Public Hospital in Lesko, Poland, Lesko, Poland

REFERENCES:
- [Background] Nuijsink M, Hop WC, Sterk PJ, Duiverman EJ, de Jongste JC. Long-term asthma treatment guided by airway hyperresponsiveness in children: a randomised controlled trial. Eur Respir J. 2007 Sep;30(3):457-66. doi: 10.1183/09031936.00111806. Epub 2007 May 30. PMID 17537770
- [Background] Lipworth BJ, Short PM, Williamson PA, Clearie KL, Fardon TC, Jackson CM. A randomized primary care trial of steroid titration against mannitol in persistent asthma: STAMINA trial. Chest. 2012 Mar;141(3):607-615. doi: 10.1378/chest.11-1748. Epub 2011 Oct 13. PMID 21998259
- [Background] Szefler SJ, Mitchell H, Sorkness CA, Gergen PJ, O'Connor GT, Morgan WJ, Kattan M, Pongracic JA, Teach SJ, Bloomberg GR, Eggleston PA, Gruchalla RS, Kercsmar CM, Liu AH, Wildfire JJ, Curry MD, Busse WW. Management of asthma based on exhaled nitric oxide in addition to guideline-based treatment for inner-city adolescents and young adults: a randomised controlled trial. Lancet. 2008 Sep 20;372(9643):1065-72. doi: 10.1016/S0140-6736(08)61448-8. PMID 18805335
- [Background] Voorend-van Bergen S, Vaessen-Verberne AA, Brackel HJ, Landstra AM, van den Berg NJ, Hop WC, de Jongste JC, Merkus PJ, Pijnenburg MW. Monitoring strategies in children with asthma: a randomised controlled trial. Thorax. 2015 Jun;70(6):543-50. doi: 10.1136/thoraxjnl-2014-206161. Epub 2015 Mar 30. PMID 25825006
- [Background] Virchow JC, Backer V, de Blay F, Kuna P, Ljorring C, Prieto JL, Villesen HH. Defining moderate asthma exacerbations in clinical trials based on ATS/ERS joint statement. Respir Med. 2015 May;109(5):547-56. doi: 10.1016/j.rmed.2015.01.012. Epub 2015 Feb 3. PMID 25676887
- [Background] Voorend-van Bergen S, Vaessen-Verberne AA, Landstra AM, Brackel HJ, van den Berg NJ, Caudri D, de Jongste JC, Merkus PJ, Pijnenburg MW. Monitoring childhood asthma: web-based diaries and the asthma control test. J Allergy Clin Immunol. 2014 Jun;133(6):1599-605.e2. doi: 10.1016/j.jaci.2013.10.005. Epub 2013 Nov 28. PMID 24290276
- [Background] Nuijsink M, De Jongste JC, Pijnenburg MW. Will symptom-based therapy be effective for treating asthma in children? Curr Allergy Asthma Rep. 2013 Oct;13(5):421-6. doi: 10.1007/s11882-013-0364-x. PMID 23775350
- [Background] Moeller A, Carlsen KH, Sly PD, Baraldi E, Piacentini G, Pavord I, Lex C, Saglani S; ERS Task Force Monitoring Asthma in Children. Monitoring asthma in childhood: lung function, bronchial responsiveness and inflammation. Eur Respir Rev. 2015 Jun;24(136):204-15. doi: 10.1183/16000617.00003914. PMID 26028633
- See also: GINA guidelines — http://www.ginasthma.org